CLINICAL TRIAL: NCT06454851
Title: A Virtual Reality (VR) Intervention for Promoting Prosocial Behavior and Well-being in Youth Transitioning From Secondary to Tertiary Education: A Randomized Controlled Trial
Brief Title: A VR Intervention for Promoting Prosocial Behavior and Well-being in Youth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSEARS20240214005-01
Record Dates: First submitted 2024-05-28; First posted 2024-06-12 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-05

CONDITIONS: Youth

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VR Intervention group (Experimental): Participants in the intervention condition will be required to complete a 4-session gamified prosocial VR intervention program, one session a week for four consecutive weeks, each session lasts around 15-20 minutes.
  Interventions: Behavioral: Prosocial VR intervention
- Waitlist control group (Sham Comparator): Participants in the waitlist condition will be asked to continue their usual activity routines before their turn to receive the intervention.
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Prosocial VR intervention — A four-week gamified prosocial VR intervention program based on literature review and relevance to the local contexts will be developed for the proposed project. The intervention will be expanded to include four weekly sessions, each lasting between 15 to 20 minutes. Each session will depict a different daily life scenario-campus, lecture hall, canteen, and library, respectively. During each session, participants will engage in a series of tasks that incorporate elements of prosocial behavior or helping actions within the scene. These tasks are designed to be more comprehensive and interactive, ensuring that participants are fully immersed in the experience for the entire duration of the session.
  Arms: VR Intervention group
Other: No intervention — The waitlist control group will not receive the intervention during the study.
  Arms: Waitlist control group

SUMMARY:
The objective of the present project is to develop a gamified prosocial VR intervention for youth transitioning from secondary to tertiary education, and to test the effectiveness of the gamified prosocial VR intervention for promoting prosocial behavior and well-being.

DETAILED DESCRIPTION:
Targeting youth transitioning from secondary to tertiary education, the proposed project will adopt evidence-based intervention programs that use digital technologies to promote prosocial behavior and well-being, thereby supporting better intrapersonal and interpersonal development.

The investigators aim to develop a gamified prosocial VR intervention for youth transitioning from secondary to tertiary education and to test its effectiveness through a randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

* Age 15-19
* Secondary 6 to college year 1
* Can read traditional Chinese and understand Cantonese

Exclusion Criteria:

* History of photosensitive epilepsy
* Impairment of stereoscopic vision
* Balance problems

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Prosocial behavior | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Prosocialness Scale for Adults (PSA) will be used to measure prosocial behavior. Each item will be rated on a 5-point Likert scale, ranging from 1 (never/almost never true) to 5 (almost always/always true). Higher scores indicate a higher level of prosocial behavior.
Prosocial attitudes | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  Three items of prosocial attitudes will be revised from the Prosocial Orientation Questionnaire. Each item will be rated on a 6-point Likert scale, ranging from 1 (strongly disagree) to 6 (strongly agree). Higher scores indicate more positive prosocial attitudes.
Prosocial identity | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Internalization subscale of the Self Importance of Moral Identity Scale (SIMIS) will be adapted to assess the prosocial identity. Each item will be rated on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree). Higher scores indicate a higher level of Prosocial identity.
Prosocial intention | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Prosocial Behavioral Intentions Scale (PBIS) will be used to assess people's intentions to behave prosocially in the future. Each item will be rated on a 7-point Likert scale, ranging 1 (Definitely would not do this) to 7 (Definitely would do this). Higher scores indicate a higher level of prosocial intention.
Attitudes toward helping others | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Attitudes toward helping others scale (AHO) will be used to test attitudes towards helping others. Each item will be rated on a 5-point Likert scale, ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate more positive attitudes toward helping others.
Altruism | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  Two items from Preference Survey Module (PSM) will be adapted to assess altruism. For example, one item is: "Imagine the following situation: you won 1,000 Euro in a lottery. Considering your current situation, how much would you donate to charity? (Values between 0 and 1000 are allowed)". Elevated scores on this item reflect a greater degree of altruistic.
Online prosocial behavior | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Online Prosocial Behavior Scale (OPBS) will be used to measure online prosocial behavior. Each item will be rated on a 7-point Likert scale, ranging 1 (never) to 7 (always). Higher scores indicate a higher level of online prosocial behavior.
Empathy | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Single Item Trait Empathy Scale (SITES) will be used to measure empathy. This item will be rated on a 7-point Likert scale, ranging from 1 (strongly disagree) to 7 (strongly agree), with a higher score indicates a higher level of empathy.
Subjective happiness | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Subjective Happiness Scale (SHS) will be used to measure participants' subjective happiness. Each item will be rated on a 7-point Likert scale. Higher scores indicate a higher level of subjective happiness.
Life satisfaction | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Satisfaction with Life Scale (SWLS) will be used to measure life satisfaction. Each item will be rated on a 7-point Likert scale ranging from "Strongly Disagree" to "Strongly Agree. Higher scores indicate higher levels of life satisfaction.
Flourishing | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Flourishing Scale (FS) will be used to measure flourishing. Each statement is answered using a 7-point Likert scale (7 - strongly agree to 1 - strongly). Higher scores indicate a higher level of flourishing.
Self-esteem | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Rosenberg Self-esteem Scale (RSE) will be used to measure self-esteem. Each item will be rated on a 4-point Likert scale, ranging from 1 (strongly agree) to 4(strongly disagree). Higher scores indicate higher levels of self-esteem.
Affect | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Emmons Mood Indicator will used to measure affect. it measures two dimensions: Positive Affect and Negative Affect. Each item will be rated on a 7-point Likert scale, ranging from 1 (not at all) to 7 (extremely). Higher scores indicate a higher level of affect.
Mental health | Baseline (pre-intervention); immediately after the intervention (post-intervention); 1 month after intervention (follow-up)
  The Patient Health Questionnaire-4 (PHQ-4) will be used to measure mental health. Each item will be rated on a 4-point Likert scale: "0" for "not at all," "1" for "several days," "2" for "more than half the days," and "3" for "nearly every day." Higher scores suggest a higher likelihood of experiencing significant depression and anxiety symptoms.
Diary measures | Daily monitoring for four weeks during the intervention
  State prosocial behavior outcomes and well-being outcomes will be measured.

SECONDARY OUTCOMES:
Feelings in the VR | immediately after the intervention (post-intervention)
  Two items will be uesd to measure the sense of reality. Items are "I feel that the maze seemed very much like the one in the real world" and "The game scene made me feel like I was truly there".
Levels of difficulty | immediately after the intervention (post-intervention)
  Two items will be used to measure the levels of difficulty. Items are "The game is very difficult" and "The game is too difficult to operate".
Levels of interest | immediately after the intervention (post-intervention)
  Two items will be used to measure the levels of difficulty. Items are "This game is very interesting" and "I like this game".
Intervention satisfaction | immediately after the intervention (post-intervention and only in the last week)
  The Client Satisfaction Questionnaire-8 (CSQ-8) will used to test Intervention satisfaction. Each item will be rated on a 4-point Likert scale where "1" indicates the lowest degree of satisfaction and "4," the highest. Higher scores indicate higher intervention satisfaction.

OTHER OUTCOMES:
Socio-demographic variables | Baseline (pre-intervention)
  The following socio-demographic variables such as gender, age, level of education, and family income will be collected.

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia CHEN, Ph.D., Principal Investigator — The Hong Kong Polytechnic University